CLINICAL TRIAL: NCT02250391
Title: Placebo-controlled Study of NPB-06 in Patients With Portal Vein Thrombosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nihon Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NPB-06-04/C-01
Record Dates: First submitted 2014-09-20; First posted 2014-09-26 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Portal Vein Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NPB-06 (Experimental): 1,500 unit, 5 days continuous-infusion
  Interventions: Drug: NPB-06
- Placebo (Placebo Comparator): 0 unit, 5 days continuous-infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NPB-06 — 5 days continuous-infusion
  Arms: NPB-06
Drug: Placebo — 5 days continuous-infusion
  Arms: Placebo

SUMMARY:
Patients with portal vein thrombosis, who have chronic liver diseases especially liver cirrhosis associated with low levels of AT III, will receive intravenous injection of NPB-06 or placebo. The superiority of NPB-06 to placebo as anticoagulative agent will be verified in a randomized, double-blind, parallel-assignment design based on the proportion of patients obtained complete recanalization or partial recanalization of portal vein thrombosis.

The safety of NPB-06 will be evaluated based on adverse events and adverse drug reactions (ADRs) observed between administration and 21 days after administration in comparison with the placebo group.

ELIGIBILITY:
Inclusion Criteria:

Inpatients or outpatients meet the criteria (1)-(4) below will be enrolled in the study. Patients have to provide written informed consent for voluntary participation in the study.

1. Patients who the serum level of AT-III is 70% or less
2. Patients with portal vein thrombosis detected by ultrasonography
3. Patients who have more than 50% of the thrombus lumen occupancy
4. Patients who are older than 20 years at the time of consent

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study beforehand.

1. Patients with tumor embolus in portal vein
2. Patients with an ongoing hepatic intra-arterial chemotherapy such as implantable reservoir system
3. Patients with hepatocellular cancer of more than 3 cm in diameter or more than four hepatocellular cancers
4. Patients with residual or chronic portal vein thrombosis
5. Patients with advanced liver disease (Child-Pugh score 11 or more)
6. Patients with bleeding tendency
7. Patients who had an anticoagulation therapy (intravenous or subcutaneous dose) or hemostasis with an enzymatic hemostatic agent in the period between 7 days before contrast enhanced CT of pre-dose and the day acquired written informed consent
8. Patients who had an anticoagulation therapy (oral dose) in the period between 7 days before contrast enhanced CT of pre-dose and the day acquired written informed consent
9. Patients with a history of shock or hypersensitivity to NPB-06
10. Patients with inappropriate to contrast agents

    * A history of allergy of iodine or X-ray contrast agent
    * Complication of serious thyroid disease
    * Reduced renal function
11. Pregnant or lactating women, women of childbearing potential, or women who plan to become pregnant during the study
12. Patients who have received NPB-06
13. Patients who have received other investigational drugs within four months before consent or who are participating in other clinical studies
14. Patients otherwise ineligible for participation in the study in the investigator's or subinvestigator's opinion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The proportion of patients obtained complete recanalization or partial recanalization of portal vein thrombosis | an expected average of 2 weeks
  Contrast enhanced CT assessed by an independent radiologist

SECONDARY OUTCOMES:
The proportion of patients obtained complete recanalization of portal vein thrombosis | an expected average of 2 weeks
Reduction rate of portal vein thrombosis | Up to 3 weeks
Improvement of Child-Pugh score | Up to 5 weeks
Changes in laboratory values (congealing fibrinogenolysis system) | Up to 5 weeks
Adverse events and adverse drug reactions observed between administration and 21 ± 3 days after administration | Up to 5 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- Japan (5):
  - Chūbu
  - Hokkaido
  - Kanto
  - Kyushu
  - Osaka